CLINICAL TRIAL: NCT07240766
Title: Phase II Study of HRS-4642 in Combination With Nimotuzumab and Chemotherapy for Subjects With Borderline Resectable Pancreatic Cancer With KRAS G12D Mutation
Brief Title: HRS-4642 in Combination With Nimotuzumab and Chemotherapy for BRPC With KRAS G12D Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Hospital President, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPT05
Record Dates: First submitted 2025-11-15; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma
Keywords: pancreatic adenocarcinoma; borderline resectable; KRAS G12D mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Perioperative Treatment with HRS-4642 in Combination with Nimotuzumab and the AG Regimen
  Interventions: Drug: HRS-4642+AG+Nimotuzumab

INTERVENTIONS:
Drug: HRS-4642+AG+Nimotuzumab — HRS-4642 Injection: 500 mg intravenous infusion on Day 1, and 1200 mg intravenous infusion on Day 8, every 3 weeks per cycle. A total of 4 cycles are planned in the neoadjuvant therapy phase, and up to a maximum of 4 cycles in the adjuvant therapy phase.
  Nimotuzumab: 400 mg on Days 1 and 8, every 3 weeks per cycle. A total of 4 cycles are planned in the neoadjuvant therapy phase, and up to a maximum of 4 cycles in the adjuvant therapy phase.
  Paclitaxel for Injection (Albumin-bound): 125 mg/m² on Days 1 and 8, every 3 weeks per cycle. A total of 4 cycles are planned in the neoadjuvant therapy phase, and up to a maximum of 4 cycles in the adjuvant therapy phase.
  Gemcitabine: 1000 mg/m² on Days 1 and 8, every 3 weeks per cycle. A total of 4 cycles are planned in the neoadjuvant therapy phase, and up to a maximum of 4 cycles in the adjuvant therapy phase.
  The recommended adjuvant treatment regimen is to continue HRS-4642 + Nimotuzumab + AG for 4 cycles.

SUMMARY:
This study is a Phase II clinical trial that plans to enroll 40 patients with borderline resectable pancreatic cancer harboring a KRAS G12D mutation, aiming to evaluate the efficacy of HRS-4642 in combination with Nimotuzumab and AG in borderline resectable pancreatic cancer. The study process includes a screening period (from the signing of the informed consent form until the first dose), a treatment period (from the first dose to the discontinuation of study treatment), and a follow-up period (safety follow-up and survival follow-up after the discontinuation of study treatment).

DETAILED DESCRIPTION:
This study is a Phase II clinical trial that plans to enroll 40 patients with borderline resectable pancreatic cancer harboring a KRAS G12D mutation, aiming to evaluate the efficacy of HRS-4642 in combination with Nimotuzumab and AG in borderline resectable pancreatic cancer. The study process includes a screening period, a treatment period, and a follow-up period.

Screening Period: The screening period for this study is 28 days. Eligible subjects who complete the screening examinations and assessments will proceed to the treatment period.

Treatment Period: Subjects who pass screening will enter the neoadjuvant therapy phase, receiving treatment with HRS-4642 in combination with Nimotuzumab and the AG regimen. The predefined administration regimen is as follows:

HRS-4642: 500 mg intravenous infusion on Day 1, and 1200 mg intravenous infusion on Day 8, every 3 weeks per cycle.

Nimotuzumab: 400 mg intravenous infusion on Days 1 and 8, every 3 weeks per cycle.

Albumin-bound paclitaxel: 125 mg/m² intravenous infusion on Days 1 and 8, every 3 weeks per cycle.

Gemcitabine: 1000 mg/m² intravenous infusion on Days 1 and 8, every 3 weeks per cycle.

Neoadjuvant therapy will consist of 4 cycles. After completing 2 cycles and 4 cycles of neoadjuvant therapy, subjects will undergo radiographic imaging for efficacy evaluation. After completing 4 cycles of neoadjuvant therapy, eligibility for radical surgery will be assessed by a Multidisciplinary Team (MDT). If assessed as eligible for radical surgery, the subject will undergo surgery within 4 weeks after completing neoadjuvant therapy.

After surgery, subjects will enter the adjuvant therapy phase. Adjuvant therapy should begin within 4 to 12 weeks after surgery. The recommended adjuvant treatment regimen is to continue HRS-4642 + Nimotuzumab + AG for 4 cycles. If a subject cannot receive HRS-4642 + Nimotuzumab + AG as adjuvant therapy, the investigator will develop an adjuvant treatment plan based on a comprehensive assessment. The adjuvant therapy phase shall not exceed 4 cycles.

If the assessment determines that radical surgery is not possible, and the subject has not experienced disease progression, the subject may continue to receive study treatment if the investigator assesses that continued treatment is likely to be beneficial.

Subjects will receive HRS-4642 in combination with Nimotuzumab and AG until radiographic disease progression, unacceptable toxicity, voluntary withdrawal, loss to follow-up/death occurs (whichever comes first).

During the treatment period, subject visits will occur on Day 1 and Day 8 of each cycle, and on Cycle 1 Day 15. Tumor imaging assessments will be performed at Cycle 3 Day 1 (±7 days) and Cycle 4 Day 21 (±7 days) (upon completion of neoadjuvant therapy). For subjects who undergo radical surgery, assessments will be performed every 12 weeks (±7 days) postoperatively. For subjects who do not undergo radical surgery, subsequent assessments will be performed every 6 weeks (±7 days) until radiographic disease progression, initiation of new anti-tumor therapy, voluntary withdrawal, loss to follow-up/death occurs (whichever comes first). If clinically indicated, imaging examinations and assessments may be performed at any time. All subjects must undergo the corresponding examinations and imaging assessments at the end-of-treatment visit (if more than 4 weeks have passed since the last assessment).

Follow-up Period: After discontinuing study treatment, subjects must return to the research center for a safety follow-up visit 30 days (±7 days) after the last dose or before starting new anti-tumor therapy. Subjects will enter the survival follow-up period after the last dose of study treatment. The investigator must conduct survival follow-ups every 2 months (±7 days) until the subject dies, is lost to follow-up, the investigator terminates the study, or other study termination criteria are met (whichever comes first). For subjects who discontinue the study for reasons other than radiographic disease progression, tumor progression follow-up should continue, including radiographic assessments per the protocol-specified frequency, until disease progression, initiation of new anti-tumor therapy, etc.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years (inclusive).
* Histopathologically confirmed pancreatic cancer (originating from the pancreatic ductal epithelium).
* Radiologically confirmed borderline resectable pancreatic cancer (according to the latest NCCN guidelines definition), with no distant metastases.
* Tumor tissue testing confirms KRAS G12D mutation.
* No prior systemic anti-tumor therapy.
* At least one evaluable lesion according to RECIST v1.1 criteria.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
* Expected survival time ≥ 3 months.
* Adequate organ function meeting the following requirements (no use of any blood components or colony-stimulating factors within 2 weeks prior to enrollment):

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
  2. Platelets ≥ 80 × 10⁹/L
  3. Hemoglobin ≥ 100 g/L
  4. Serum albumin ≥ 30 g/L
  5. Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN and ALP ≤ 2.5 × ULN
  6. Creatinine clearance ≥ 50 mL/min or Serum creatinine ≤ 1.5 × ULN (Calculation formula see section 13.3)
  7. Electrocardiogram: QTcF ≤ 450 ms (male), QTcF ≤ 470 ms (female)
  8. Cardiac ultrasound: LVEF (Left Ventricular Ejection Fraction) ≥ 50%
* Women of childbearing potential must have a negative serum pregnancy test within 7 days before enrollment, must be non-lactating, and must be willing to use adequate contraception during the trial and for 6 months after the end of treatment. For men, they must be surgically sterile or agree to use adequate contraception during the study and for 6 months after the end of treatment.
* Voluntary participation in this study and signing of informed consent, good compliance, and agreement to cooperate with follow-up.

Exclusion Criteria:

* 1. Prior Treatment:

  1. Major surgical procedure or significant traumatic injury within 4 weeks prior to enrollment, or palliative local therapy (including but not limited to palliative radiotherapy, interventional therapy) within 2 weeks prior to enrollment.
  2. Treatment with any investigational drug from another clinical study within 4 weeks prior to enrollment, except for participation in an observational (non-interventional) clinical study or the follow-up phase of an interventional study.
  3. Use of strong inhibitors or inducers of hepatic drug-metabolizing enzymes CYP3A4 or CYP2C8 within 14 days prior to enrollment.
* 2. Acute or chronic pancreatitis requiring clinical intervention.
* 3. History or presence of symptoms/signs of gastrointestinal obstruction within 6 months prior to the start of study treatment. Subjects may be screened if they have undergone surgical procedure resulting in complete resolution of the obstruction.
* 4. Third-space fluid accumulation (e.g., significant pleural effusion, ascites, etc.) that is unstable (unable to remain stable without intervention after drainage removal) within 2 weeks prior to enrollment. Subjects with only small amounts of fluid visible on imaging and without clinical symptoms may be enrolled.
* 5. Severe infection within 4 weeks prior to enrollment, such as severe pneumonia, bacteremia, or infectious complications requiring hospitalization; Unexplained fever >38.5°C within 2 weeks prior to enrollment (subjects with fever judged by the investigator to be due to the tumor may be enrolled); Presence of signs/symptoms of infection requiring intravenous antibiotic therapy within 2 weeks prior to enrollment (excluding prophylactic antibiotic use).
* 6. Severe cardiovascular and cerebrovascular diseases:

  1. Important arterial/venous thrombotic events within 6 months prior to enrollment, such as cerebrovascular accident (including cerebral hemorrhage, cerebral infarction), deep vein thrombosis (excluding muscular venous thrombosis not requiring anticoagulation), and pulmonary embolism.
  2. Poorly controlled cardiac symptoms or diseases, such as:

     1. Myocardial infarction within 6 months.
     2. Unstable angina.
     3. Heart failure of NYHA class II or above.
     4. Subjects with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
* 7. Patients with known or suspected interstitial lung disease, with the exception of interstitial changes visible only on imaging without clinical symptoms.
* 8. History of definite neurological or psychiatric disorders, including epilepsy and dementia.
* 9. Presence of non-healed wounds (severe, non-healing, or dehisced) or unhealed fractures.
* 10. Adverse events from prior anti-cancer therapy have not recovered to NCI-CTCAE grade ≤1 (except for alopecia and parameters already specified in the inclusion criteria; except for AEs judged by the investigator as not affecting study drug administration).
* 11. History of other malignant tumors within 5 years prior to enrollment, except for those with low risk of metastasis and death: adequately treated carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, etc.
* 12. Concurrent active Hepatitis B (if HBsAg positive, HBV DNA must be tested; HBV DNA <2000 IU/mL is required for enrollment and the subject must receive standard antiviral therapy during the study), Hepatitis C (HCV antibody positive and HCV-RNA above the lower limit of detection of the assay). Known history of acquired immunodeficiency syndrome or positive HIV test. Active syphilis infection. Active tuberculosis or history of active tuberculosis infection within 48 weeks prior to screening, regardless of treatment.
* 13. Known allergy to any component of HRS-4642; history of allergy to Nimotuzumab, other monoclonal antibody/fusion protein drugs, albumin-bound paclitaxel, or gemcitabine.
* 14. Any other condition that, in the judgment of the investigator, may affect the study results or lead to the premature termination of the study, such as alcoholism, drug abuse, other serious concomitant diseases (including psychiatric disorders) requiring treatment, severely abnormal laboratory test values, family or social factors, and other circumstances that may affect patient safety or reliability of data collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
12-month Event-Free Survival (EFS) rate | Up to one year
  The proportion of patients who had tumor progression, tumor recurrence (local, regional or distant) or death within 1 year after surgery, whichever occurred first

SECONDARY OUTCOMES:
Event Free Survival, EFS | Up to 2 years
  From treatment to the date of the first documented tumor progression, tumor into recurrence or death from any cause, whichever occurred first
Surgical resection rate | Up to 1 year
  The proportion of patients who receive the radical resection
R0 resection rate | Up to 1 year
  R0 resection rate is the percentage of patients who undergo a surgical procedure where the surgeon successfully removes the entire visible tumor and a microscopic examination confirms that no cancer cells are left at the edges (margins) of the removed tissue.
Pathological Complete Response (pCR) Rate | Up to 1 year
  The percentage of patients who, after pre-surgical (neoadjuvant) therapy, have no viable cancer cells detected in the tumor tissue and lymph nodes that are removed during subsequent surgery when examined under a microscope by a pathologist.
Major Pathological Response (MPR) Rate | Up to 1 year
  The percentage of patients who, after neoadjuvant therapy, have only a minimal amount of viable tumor remaining in the resected specimen. This is typically defined as ≤10%
Objective Response Rate (ORR) | Up to 2 years
  The proportion of patients whose tumor shrinks (responds) by a predefined amount from its baseline size for a minimum period of time. It includes two categories of response:
  Complete Response (CR): The disappearance of all target tumors. Partial Response (PR): A specified minimum decrease (e.g., 30%) in the sum of the diameters of the target tumors.
Disease Control Rate (DCR) | Up to 2 yeas
  The proportion of patients who have achieved a best response of either Stable Disease (SD), Partial Response (PR), or Complete Response (CR). It essentially measures the treatment's ability to stop the cancer from growing.
Overall Survival (OS) | Up to 3 yeas.
  The length of time from a defined point in a study (e.g., date of randomization or start of treatment) until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Patient Privacy and Ethical Compliance: The dataset contains detailed, sensitive clinical information. Ensuring complete and irreversible anonymization of participants is challenging, and sharing IPD could potentially compromise patient confidentiality and violate the ethical commitments made to participants and the approving IRB. For researchers interested in specific analytical outcomes or validated findings, the corresponding author may be contacted to discuss the possibility of collaborative re-analysis where feasible and subject to a formal data sharing agreement.